CLINICAL TRIAL: NCT01695811
Title: Femtosecond Laser-Assisted Keratoplasty
Acronym: FLAK
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Shahzad Mian, Professor, Department of Ophthalmology, University of Michigan
Other Study IDs: FLAK-15615
Record Dates: First submitted 2012-09-27; First posted 2012-09-28 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Keratoconus
Keywords: Keratoconus, PKP, femtosecond laser assisted keratoplasty
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FLAK: FLAK
- PKP: Retrospective

SUMMARY:
The purpose of this study will be to determine optimal surgical technique for performing FLAK including laser parameters, keratoplasty shape and suture technique in order to standardize surgical technique and to collect safety and efficacy data. This will be compared to data of patients with full thickness PKP to measure visual outcomes, refraction, astigmatism, surgical methods and wound healing.

DETAILED DESCRIPTION:
FLAK Instrument: The Femtosecond Laser (IntraLase Corporation, Irvine, CA) is a focusable infrared laser, similar to the more familiar neodymium-yttrium-aluminum-garnet (YAG) laser, but uses shorter pulses in the hundred-femtosecond (100 X 10-15 seconds) duration range. There is minimal postoperative inflammation and collateral tissue damage.

Subjects: We will be enrolling subjects 18 years or older that need keratoplasty based on clinical findings. Subjects will be enrolled regardless of race or gender on a first come first serve basis. Subjects will be recruited from the physicians own clinic.

PKP Subjects: We will do a retrospective chart review on subjects who have undergone traditional PKP. FLAK eyes will be age and gender matched to these PKP eyes to compare visual outcomes, wound healing and complications.

ELIGIBILITY:
Inclusion Criteria:

1. Corneal opacification.
2. Reduced ETDRS-measured, best corrected, distance visual acuity to 20/40 or worse.
3. Ability to participate in follow-up visits..

Exclusion Criteria:

1. Corneal opacification adequately dense to obscure visualization of iris.
2. ETDRS-measured, best-corrected, distance visual acuity of 20/30 or better.
3. Corneal thickness greater than 1200 µm at the 9 mm peripheral zone.
4. Severe corneal thinning including descemetocoele with impending corneal rupture.
5. Prior PKP or incisional surgery that may provide a potential space into which the gas produced by the procedure can escape.
6. Poor visual potential in the non-study eye (VA of 20/100 or less, without potential for improvement by the examining ophthalmologist's judgment).
7. History of glaucoma, including steroid response rise in intraocular pressure.
8. Active intraocular inflammation or infection.
9. Age 18 or younger (consideration will be given to an upper age limit).
10. Unable to return for scheduled follow-up examinations.
11. Other medical condition(s) that will likely prevent long term follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects indicated for corneal transplant surgery
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2007-11; Primary Completion 2012-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Surgical outcomes | 1 day, 1 week, 1, 3, 6, 12, 18 and 24 months
  Wound healing, surgical complications, visual function and endothelial layer assessment